CLINICAL TRIAL: NCT01453777
Title: An Open-label, Non-Randomized, Multi-Center Study to Assess the Safety and Effects of Autologous Adipose-Derived Stromal Cells Delivered Via Catheter Into the Internal Carotid Artery and Intravenously in Patients With Diffuse Lesions in the Brain
Brief Title: Safety and Effects of Autologous Adipose-Derived Stromal Cells in Patients With Diffuse Lesions in the Brain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Ageless Regenerative Institute (Industry)
Collaborators: Instituto de Medicina Regenerativa (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADI-ME-DL-001
Record Dates: First submitted 2011-10-03; First posted 2011-10-18 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-03

CONDITIONS: Brain Lesion (General)
Keywords: diffuse brain lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: harvesting and implantation of adipose derived stem cells — Adipose-Derived Stem cells will be derived from the patient's fat tissue. Liposuction using local anesthesia and syringe collection will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells. The cells will be delivered via catheter into the internal carotid artery and intravenously.

SUMMARY:
The intent of this clinical study is to answer the questions:

1. Is the proposed treatment safe
2. Is treatment effective in improving the disease pathology of patients with diffuse brain lesions and clinical outcomes.

DETAILED DESCRIPTION:
This will be an open-label, non-randomized multi-center patient sponsored study of Adipose-Derived Stromal Cells (ASC) implantation using a catheter delivery system. ASCs will be derived from the patient's adipose-derived tissue. Liposuction using local anesthesia and syringe collection will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells. The cells will be delivered via catheter into the internal carotid artery and intravenously.

ELIGIBILITY:
Inclusion Criteria:

* Males and Females between Age 18 and 80 years.
* Patient with current diagnosis of Diffuse Brain Lesions with cognitive and/or functional impairment
* MRI not showing gross atrophy or any other pathology of brain.
* Up to date on all age and gender appropriate cancer screening per American Cancer Society

Exclusion Criteria:

* Contraindication for MRI
* General medical contraindications for minor surgery or angiography
* Females who are pregnant or nursing or females of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Active infectious disease. Patients known to have tested positive will have an expert consulted as to patient eligibility based on the patient's infectious status
* Any illness which, in the Investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* Patients on chronic immunosuppressive transplant therapy
* Systolic blood pressure (supine) ≤90 mmHg;
* Resting heart rate > 100 bpm;
* Active clinical infection within one week of enrollment.
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* History of cancer (other than non-melanoma skin cancer or in-situ cervical cancer) in the last five years.
* Unwilling and/or not able to give written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in standardized Gross Motor Function Measure evaluation compared to baseline | 3 months
Number of participants with adverse events | up to 6 months
  The safety of adipose-derived stem cell injection will be evaluated by assessment of the frequency and nature of adverse events occurring during the study injection and up to the 6-month period following treatment.
Improved cognitive function as measured by the mini mental state exam | 3 months
Improvement in standardized Gross Motor Function Measure evaluation compared to baseline | 6 months
Improved cognitive function as measured by the mini mental state exam compared to baseline | 6 months
Reduced depressive symptoms measured by the Beck Depression Inventory compared to baseline | 3 months
Reduced depressive symptoms measured by the Beck Depression Inventory compared to baseline | 6 months

SECONDARY OUTCOMES:
number of brain lesions by MRI compared to baseline | 3 months
Improved quality of life scores compared to baseline | 3 months
Improved quality of life scores compared to baseline | 6 months
number of brain lesions by MRI compared to baseline | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Victor D Morales, MD, Principal Investigator — Instituto de Medicina Regenerativa; Clemente Zuñiga, md, Principal Investigator — Instituto de Medicina Regenerativa
Locations (1):
- Hospital Angeles, Tijuana, Estado de Baja California, Mexico